CLINICAL TRIAL: NCT03111056
Title: Web-Based Treatment of Heavy Drinking Among Women With a History of Sexual Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Cynthia Stappenbeck, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001028
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Sexual Assault; Heavy Drinking

STUDY DESIGN:
Masking Description: The intervention and assessments are all completed online and therefore masking is not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Intervention (Experimental): In an effort to reduce heavy drinking, participants will be asked to complete a daily monitoring assessment each morning for 14 days. Based on their responses, they will be provided a coping skill to either directly address their alcohol use or attempt to improve their emotion regulation and distress tolerance skills.
  Interventions: Behavioral: Alc-ERDT
- Assessment Only Control (No Intervention): Participants will be asked to complete only the daily monitoring assessment each morning for 14 days.

INTERVENTIONS:
Behavioral: Alc-ERDT — Web-based cognitive behavioral skills-based alcohol intervention that incorporates emotion regulation and distress tolerance skills
  Arms: Web-Based Intervention

SUMMARY:
The goal of this study is to empirically evaluate a web-based intervention to reduce heavy drinking among college women with a history of sexual assault who display elevated levels of psychological distress. College women with a history of sexual assault often report more heavy drinking and psychological distress than women without a history of assault. Moreover, women with assault histories often have difficulty regulating their emotions and tolerating distress which can lead to a pattern of drinking to cope distress. Trauma exposure, negative mood, and poor coping strategies have been associated with poor treatment outcomes and relapse following alcohol treatment. Incorporating distress tolerance and emotion regulation skills with an alcohol intervention may enhance treatment effects among women with a history of sexual assault by decreasing their motivation to drink to cope with depression or anxiety and by building adaptive coping strategies. Therefore, the web-based intervention will include cognitive behavioral skills for reducing alcohol consumption and incorporate emotion regulation and distress tolerance skills from Dialectical Behavior Therapy.

DETAILED DESCRIPTION:
For the small randomized controlled trial, heavy drinking college women with a history of sexual assault will be recruited and randomized to receive the intervention or an assessment only control. Online surveys will be administered at baseline, and post-treatment as well as 1-month and 6-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment at the University of Washington,
* female,
* 18 or older,
* lifetime history of sexual assault (defined as unwanted attempted or completed oral, vaginal, or anal penetration but excluding unwanted sexual contact only),
* at least 2 instances of heavy episodic drinking (defined as 4 or more drinks in 2 hours) in the past 30 days,
* average consumption equal or greater than 7 drinks per week in the past 30 days.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified as female
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Changes in Daily Drinking Questionnaire | Baseline, Immediately upon completion of the intervention, 1-month and 6-month follow-up
  Assesses typical alcohol consumption over the course of a typical week in the past month

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Stappenbeck, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No